CLINICAL TRIAL: NCT01527045
Title: Donor Statin Treatment for Prevention of Severe Acute GVHD After Nonmyeloablative Hematopoietic Cell Transplantation
Brief Title: Donor Atorvastatin Treatment in Preventing Severe Acute GVHD After Nonmyeloablative Peripheral Blood Stem Cell Transplant in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2546.00; NCI-2011-03828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2546.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; Blasts Under 5 Percent of Bone Marrow Nucleated Cells; Chronic Lymphocytic Leukemia; Loss of Chromosome 17p; Myelodysplastic/Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Aggressive Adult Non-Hodgkin Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma; Recurrent Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Non-Hodgkin; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma, Mantle-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Atorvastatin; Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (donor statin treatment) (Experimental): See Detailed Description
  Interventions: Drug: Atorvastatin Calcium; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Atorvastatin Calcium — Given PO
  Other Names: ATORVASTATIN CALCIUM TRIHYDRATE; CI-981; Lipitor
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo nonmyeloablative allogeneic PBSC transplant
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo nonmyeloablative allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well donor atorvastatin treatment works in preventing severe graft-versus-host disease (GVHD) after nonmyeloablative peripheral blood stem cell (PBSC) transplant in patients with hematological malignancies. Giving low doses of chemotherapy, such as fludarabine phosphate, before a donor PBSC transplantation slows the growth of cancer cells and may also prevent the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also cause an immune response against the body's normal cells (GVHD). Giving atorvastatin to the donor before transplant may prevent severe GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether 2 weeks of donor statin treatment reduces the risk of severe acute GVHD.

SECONDARY OBJECTIVES:

I. To assess whether 2 weeks of statin treatment of normal PBSC donors is feasible, tolerable and safe.

OUTLINE:

DONOR: Donors receive atorvastatin orally (PO) once daily (QD) beginning on day -14 and continuing until the last day of stem cell collection.

NONMYELOABLATIVE PREPARATIVE REGIMEN: If the patient is enrolled on an investigational nonmyeloablative hematopoietic cell transplant (HCT) protocol or a treatment plan that uses a nonmyeloablative preparative regimen with postgrafting cyclosporine (CSP) that does not use acute GVHD as its primary endpoint, the preparative regimen and immunosuppression after transplant will be according to respective protocol or treatment plan (Protocol 2546 serves as adjunct protocol).

If the patient is not enrolled on an investigational nonmyeloablative HCT protocol or a treatment plan that uses a nonmyeloablative preparative regimen, Protocol 2546 serves as an independent primary treatment protocol. The preparative regimen and immunosuppression after transplant is as follows:

Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 (except for patients who had prior autologous HCT or equivalent high-dose therapy without HCT) and undergo low-dose total body irradiation (TBI) on day 0.

TRANSPLANT: Patients undergo donor PBSC transplant on day 0.

POST-GRAFTING IMMUNOSUPPRESSION: Patients receive CSP PO twice daily (BID) on days -3 to 56 with taper to day 180. Patients also receive mycophenolate mofetil (MMF) PO BID or IV every 12 hours on days 0-27.

After completion of study treatment, patients are followed up at 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

IF PROTOCOL 2546 SERVES AS AN ADJUNCT PROTOCOL, THE PATIENTS ONLY NEEDS TO MEET INCLUSION CRITERIA 1 THROUGH 5A

* Availability of human leukocyte antigen (HLA)-identical sibling donor
* Transplantation with PBSC
* CSP-based postgrafting immunosuppression
* Willingness to give informed consent
* Patient is enrolled on an investigational nonmyeloablative HCT protocol or a nonmyeloablative treatment plan with postgrafting CSP that does not use acute GVHD as its primary endpoint (protocol 2546 serves as adjunct protocol); OR
* Patient is not enrolled on an investigational nonmyeloablative HCT protocol, in which case protocol 2546 serves as an independent primary treatment protocol and the patient must meet the following inclusion and exclusion criteria:
* Patients must have a hematologic malignancy treatable by nonmyeloablative HCT; the following diseases will be permitted although other diagnoses can be considered if approved by Patient Care Conference (PCC) and the principal investigator:
* Aggressive non-Hodgkin lymphomas (NHL) and other histologies such as diffuse large B-cell NHL - not eligible for autologous HCT, not eligible for high-dose allogeneic HCT, or after failed autologous HCT
* Mantle-cell NHL - may be treated in first complete remission (CR); (diagnostic lumbar puncture [LP] required pre-transplant)
* Low grade NHL - with < 6 month duration of CR between courses of conventional therapy
* Chronic lymphocytic leukemia (CLL) - must have either:

  * Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine phosphate (FLU) (or another nucleoside analog) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog)
  * Failed FLU-cyclophosphamide (CY)-Rituximab (FCR) combination chemotherapy at any time point; or
  * Have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in 1st CR
  * Patients with a diagnosis of CLL (or small lymphocytic lymphoma) that progresses to prolymphocytic leukemia (PLL); or
  * Patients with T-cell CLL or PLL
* Hodgkin lymphoma - must have received and failed frontline therapy
* Multiple myeloma - must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
* Acute myeloid leukemia (AML) - must have < 5% marrow blasts at the time of transplant
* Acute lymphocytic leukemia (ALL) - must have < 5% marrow blasts at the time of transplant
* Chronic myeloid leukemia (CML) - Patients will be accepted if they have shown intolerance to tyrosine kinase inhibitors or are beyond first chronic phase (CP1) and if they have received previous myelosuppressive chemotherapy or HCT, and have < 5% marrow blasts at time of transplant
* Myelodysplasia (MDS)/myeloproliferative syndrome (MPS) - Patients must have < 5% marrow blasts at time of transplant
* Waldenstrom's macroglobulinemia - must have failed 2 courses of therapy
* Patients < 12 years of age must be approved by the principal investigator and by a relevant patient review committee, such as the Fred Hutchinson Cancer Research Center (FHCRC) Patient Care Conference (PCC)
* Patients must have either relapsed after previous high-dose chemotherapy and autologous or allogeneic HCT, or else be ineligible for such an approach due to age, failure to mobilize sufficient hematopoietic stem cells, medical comorbidities, or patient refusal
* Patients who refuse to be treated on a conventional autologous or allogeneic HCT protocol
* DONOR: Age >= 18 years
* DONOR: HLA genotypically identical sibling
* DONOR: Willingness to give informed consent

Exclusion Criteria:

IF PROTOCOL 2546 SERVES AS AN ADJUNCT PROTOCOL, THE PATIENT ONLY NEEDS TO MEET EXCLUSION CRITERIA 1 THROUGH 3

* Myeloablative preparative regimen
* Participation in an investigational study that has acute GVHD as the primary endpoint
* The allogeneic PBSC donor has a contraindication to statin treatment
* Patients eligible for and willing to receive potentially curative high-dose chemotherapy and autologous HCT
* Cardiac ejection fraction < 30% on multi gated acquisition scan (MUGA) scan or cardiac echocardiogram (echo) or active symptomatic coronary artery disease; patients with cardiac disease should be evaluated with appropriate cardiac studies and/or cardiology consultation as clinically indicated
* Corrected diffusion capacity of the lung for carbon monoxide (DLCO) < 40% of predicted, total lung capacity (TLC) < 30% of predicted, forced expiratory volume in one second (FEV1) < 30% of predicted, or receiving continuous supplementary oxygen
* Patients with clinical or laboratory evidence of liver disease should be evaluated in conjunction with the gastrointestinal (GI) consult service for the cause of the liver disease, its clinical severity, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, refractory ascites related to portal hypertension, bacterial or fungal liver abscess, chronic viral hepatitis with total serum bilirubin > 3mg/dl, or actively symptomatic biliary disease
* Patients with renal failure are eligible; however, patients with pre-existing renal insufficiency will likely have further compromise in renal function and may require dialysis
* Patients who are seropositive for human immunodeficiency virus (HIV)
* Women who are pregnant or breast-feeding
* Fertile men or women unwilling to use contraception during HCT and for 12 months afterward
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Karnofsky score < 60 for adult patients
* Lansky-play performance score < 50 for pediatric patients
* Patients with fungal pneumonia with radiological progression after receipt of amphotericin formulation or mold-active azoles for greater than 1 month
* DONOR: Age < 18 years
* DONOR: History of liver disease; a donor with a history of liver disease would be eligible if the serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) are < 2 times upper limit of normal (ULN)
* DONOR: History of myopathy
* DONOR: Hypersensitivity to atorvastatin
* DONOR: Pregnancy
* DONOR: Nursing mother
* DONOR: Current serious systemic illness
* DONOR: Concurrent treatment with strong inhibitors of hepatic CYP 3A4 (i.e. clarithromycin, erythromycin, protease inhibitors, azole antifungals)
* DONOR: Failure to meet local criteria for stem cell donation
* DONOR: Total creatinine kinase > 2 times the ULN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-09-25 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary - Reg A (Flu/TBI): NONMYELOABLATIVE PREPARATIVE REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 (except for patients who had prior autologous HCT or equivalent high-dose therapy without HCT) and undergo low-dose total body irradiation (TBI) on day 0.
  TRANSPLANT: Patients undergo donor PBSC transplant on day 0.
  POST-GRAFTING IMMUNOSUPPRESSION: Patients receive CSP PO twice daily (BID) on days -3 to 56 with taper to day 180. Patients also receive mycophenolate mofetil (MMF) PO BID or IV every 12 hours on days 0-27.
- Primary - Reg B (TBI Alone): NONMYELOABLATIVE PREPARATIVE REGIMEN: Patients will undergo low-dose total body irradiation (TBI) on day 0.
  TRANSPLANT: Patients undergo donor PBSC transplant on day 0.
  POST-GRAFTING IMMUNOSUPPRESSION: Patients receive CSP PO twice daily (BID) on days -3 to 56 with taper to day 180. Patients also receive mycophenolate mofetil (MMF) PO BID or IV every 12 hours on days 0-27.
- Adjunct: NONMYELOABLATIVE PREPARATIVE REGIMEN: The preparative regimen and immunosuppression after transplant will be according to respective protocol or treatment plan.
  POST-GRAFTING IMMUNOSUPPRESSION: Patients receive CSP PO twice daily (BID) on days -3 to 56 with taper to day 180. Patients also receive mycophenolate mofetil (MMF) PO BID or IV every 12 hours on days 0-27.
Period: Overall Study
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Started | 30 | 5 | 12
Completed | 29 | 5 | 12
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct | Total
Number analyzed (Participants) | 30 | 5 | 12 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 9 | 26
  >=65 years | 17 | 1 | 3 | 21
Age, Continuous [Median (Full Range); unit: years] | 65.4 [26.8 to 79.5] | 54 [35 to 66.9] | 62.35 [53.6 to 74.5] | 64.1 [26.8 to 79.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 3 | 16
  Male | 20 | 2 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 5 | 12 | 46
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 25 | 4 | 10 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 5 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade III-IV Acute Graft-versus-host Disease (GVHD) Post-transplant
Description: Number of patients who developed acute GVHD post allogeneic transplant.
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: 100 days post-transplant
Population: One subject on Reg A aborted transplant during conditioning due to donor related medical issue and subsequently went on to transplant on a different study. This subject was counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 2 | 0 | 0

2. Secondary Outcome: Number of Patients With Grades II-IV Acute Graft-versus-host-disease (GVHD)
Description: as for outcome 1
Time Frame: 100 days post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 15 | 2 | 6

3. Secondary Outcome: Number of Patients Requiring Secondary Systemic Immunosuppressive Therapy
Description: Number of patients requiring systemic immunosuppressive therapy other than those used for prophylaxis and initial therapy.
Time Frame: 1 Year post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 23 | 3 | 4

4. Secondary Outcome: Number of Patients With Chronic Extensive GVHD
Description: Number of patients who developed chronic extensive GVHD post-transplant. The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD. Patients were evaluated as described in the National Institutes of Health (NIH) consensus project guidelines.
Time Frame: 1 Year post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 8 | 1 | 5

5. Secondary Outcome: Number of Patients With Recurrent or Progressive Malignancy
Description: CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever greater than 38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  AML, ALL, MDS >5% marrow blasts by morphologic or flow cytometric, or appearance of extramedullary disease.
  CLL ≥1 of: Physical exam/Imaging studies (nodes, liver, and/or spleen) ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or number of plasmacytomas or lytic bone lesions.
Time Frame: 1 Year post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 7 | 4 | 3

6. Secondary Outcome: Number of Non-relapse Mortalities
Description: Number of patients who died without relapsed/progressive disease.
Time Frame: 1 Year post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 4 | 1 | 0

7. Secondary Outcome: Number of Patients Surviving Overall
Description: Number of patients surviving overall post-transplant
Time Frame: 1 Year post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 29 | 5 | 12
Participants | 21 | 3 | 9

8. Secondary Outcome: Number of Donors Discontinuing Atorvastatin Due to Toxicity
Description: The number of donors who prematurely discontinue atorvastatin therapy due to toxicity. Donors will be assessed for the following events:
  * Musculoskeletal and connective tissue disorders: grade 2-5
  * Hepatobiliary disorders: grade 2-5
  * Other unexpected events thought related to the use of atorvastatin; grade 2-5
  In cases where the NCI criteria do not apply, intensity will be defined as:
  * Mild: awareness of symptom or sign, but easily tolerated
  * Moderate: discomfort is enough to cause interference with normal activities
  * Severe: inability to perform normal daily activities
  * Life threatening: immediate risk of death from the reaction as it occurred
Time Frame: Prior to stem cell collection
Measure: Count of Participants; unit: Participants
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
Number analyzed (Participants) | 30 | 5 | 12
Participants | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200; All-Cause Mortality: Conditioning through 1 Year.
Arm/Group | Primary - Reg A (Flu/TBI) | Primary - Reg B (TBI Alone) | Adjunct
All-Cause Mortality (participants affected / at risk) | 8/29 | 2/5 | 3/12
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 6/29 | 1/5 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary - Reg A (Flu/TBI) (N=29) | Primary - Reg B (TBI Alone) (N=5) | Adjunct (N=12)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary - Reg A (Flu/TBI) (N=29) | Primary - Reg B (TBI Alone) (N=5) | Adjunct (N=12)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT01527045/Prot_SAP_000.pdf